CLINICAL TRIAL: NCT00476879
Title: Growth Hormone During Fasting. Signaltransduktion in Muscle and Adipose Tissue, Consequence of Growth Hormone Receptor Antagonist, Quantification of Intrahepatic Lipid Content Based on MR Scanning
Brief Title: Growth Hormone During Fasting.Signaltransduktion in Muscle and Adipose Tissue and Changes in Intrahepatic Lipid Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Pfizer (Industry)
Responsible Party: Jens Otto Lunde Jorgensen, Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 090600-deleted
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Metabolism; Fatty Liver
Keywords: Growth hormone; Fasting; Signaltransduction; fatty liver; insulin sensitivity; forearm model; protein metabolism; respiratory quotient
MeSH Terms: conditions — Fatty Liver; Fasting; Insulin Resistance | interventions — Human Growth Hormone; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 12 hours of fasting and a GH bolus
  Interventions: Drug: Somatropin and pegvisomant
- 2 (Experimental): 36 hours of fasting and a GH bolus
  Interventions: Drug: Somatropin and pegvisomant
- 3 (Experimental): 36 hours of fasting and Pegvisomant
  Interventions: Drug: Somatropin and pegvisomant
- 4 (Experimental): 36 hours of fasting and NaCl injection
  Interventions: Drug: Somatropin and pegvisomant

INTERVENTIONS:
Drug: Somatropin and pegvisomant — Somatropin are given intravenous, 0.5mg pegvisomant are given subcutaneous, 15 mg NaCl are given subcutaneous, 2 ml

SUMMARY:
The purpose of this study is to examine the effects of growth hormone during fasting in healthy lean men.

DETAILED DESCRIPTION:
During fasting the human body is known to metabolize relatively large amounts of fat, in the expense of proteins and glucose. Partly this shift in metabolism is caused by increasing GH secretion, but exactly how growth hormone exerts these effects remains to be further investigated.

10 healthy lean young men are studied at 4 different occasions in a randomized single-blinded cross-over study. 1: after 12 hours of fasting + GH bolus, 2: after 36 hours of fasting + GH bolus, 3: after 36 hours + saline, 4: after 36 hours of fasting + Somavert.

Aim:

* to study the signal transduction in muscle and fat tissue
* to study the metabolism during fasting
* to study the intrahepatic fat content using magnetic resonance techniques

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* age 20 - 40 years of age
* BMI 20 -25

Exclusion Criteria:

* uses any medication
* drinks more than 21 units of alcohol per
* is claustrophobic
* carries any magnetic devices

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
changes in intrahepatic lipid content | 12 and 36 hours of fasting. respectively
changes in intracellular signaling during fasting | 36 hours
changes in respiratory quotient | 36 hours of fasting
metabolism | 36 hours of fasting
insulin sensitivity | 36 hours of fasting
forearm metabolism | 36 hours of fasting

SECONDARY OUTCOMES:
changes in FFA | 36 hours of fasting
Changes in grelin | 36 hours of fasting
changes in leptin, adiponektin, cortisol, catecholamine, glucagon, carbamide, palmitate | 36 hours of fasting

CONTACTS AND LOCATIONS:
Overall Officials: Louise Moller, MD, Principal Investigator — Medical department M, Aarhus Sygehus, Norrebrogade 44, 8000 Aarhus, Denmark
Locations (1):
- Medical department M, Arhus Sygehus, Region midtjylland, Aarhus, Denmark

REFERENCES:
- [Derived] Moller L, Norrelund H, Jessen N, Flyvbjerg A, Pedersen SB, Gaylinn BD, Liu J, Thorner MO, Moller N, Lunde Jorgensen JO. Impact of growth hormone receptor blockade on substrate metabolism during fasting in healthy subjects. J Clin Endocrinol Metab. 2009 Nov;94(11):4524-32. doi: 10.1210/jc.2009-0381. Epub 2009 Oct 9. PMID 19820031